CLINICAL TRIAL: NCT00308815
Title: Comparison of Manual Cardiopulmonary Resuscitation (CPR) Versus Automatic CPR Machine on the CPR Performance for Out-of-Hospital Cardiac Arrest During Ambulance Transport.
Brief Title: Comparison of Manual Cardiopulmonary Resuscitation (CPR) Versus Automatic CPR Machine During Ambulance Transport.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 9361701098
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Last update posted 2006-03-30 (Estimated); Status verified 2004-10

CONDITIONS: Cardiac Arrest; Cardiopulmonary Resuscitation
Keywords: Resuscitation; Out-of-hospital cardiac arrest; cardiac arrest; CPR
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

INTERVENTIONS:
Device: Automatic CPR machine

SUMMARY:
This is a randomized controlled prospective study which assigned patient to receive manual CPR or automatic CPR machine use. The quality and efficacy between manual CPR and machine CPR will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Non-traumatic out-of-hospital cardiac arrest patient in Taipei distric
* Patients sent to National Taiwan University Hospital (NTUH) through Jhongsiao Emergency medical service (EMS) team

Exclusion Criteria:

* Younger than 15 years old
* Traumatic cardia arrest
* Patients not sent to NTUH by Jhongsiao EMS team

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2005-01

PRIMARY OUTCOMES:
Quality of CPR

SECONDARY OUTCOMES:
End-tidal CO2 on arrival at ER
Recovery of spontaneous circulation (ROSC) rate
Survival rate at 1hr, 24hr, and discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chu Chiang, M.D., Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan